CLINICAL TRIAL: NCT00633425
Title: Continuous Glucose Monitoring System (CGMS) in Type 2 Diabetic Patients Inadequately Controlled by Metformine Monotherapy; Analyze of Glycemic Profile Before and After Association of Glimepiride
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE490B_4001
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — glimepiride

INTERVENTIONS:
Drug: GLIMEPIRIDE

SUMMARY:
Analyse the glucose profile, based on continuous glucose monitoring by CGMS, in type 2 diabetics inadequately controlled by metformin, before and after the addition of Glimepiride.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 35 to 70 years
* Having given their consent
* Type 2 diabetics (HBA1c greater than 6.5%
* Fasting glycaemia greater than 1.40 g/l) not controlled by Metformin for at least 6 weeks.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2002-10; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Change in interstitial glucose levels between the observation and maintenance phases. | The mean of 24 variations in average hourly glucose readings recorded by CGMS.

SECONDARY OUTCOMES:
HbA1c and fasting blood glucose levels. | Measured in the observation and maintenance phases, and change between the two phases.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Billon, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France